CLINICAL TRIAL: NCT05371275
Title: Phase II Safety Single-arm Study of CDK4/6 Inhibition With Palbociclib in Hospitalized, Moderate COVID-19 Cases to Prevent Thromboinflammation
Acronym: CDK6COV
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was withdrawn due to challenges in patient enrollment
Sponsor: biotx.ai GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BXAI-001; 2021-006770-24 (EudraCT Number)
Record Dates: First submitted 2022-04-26; First posted 2022-05-12 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: COVID-19
Keywords: COVID-19; moderate; hospitalized; Palbociclib; CDK4/6 inhibition
MeSH Terms: conditions — COVID-19; Lymphoma, Follicular | interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Palbociclib (Experimental): 125 mg of palbociclib once daily for 21 consecutive days
  Interventions: Drug: Palbociclib

INTERVENTIONS:
Drug: Palbociclib — 125 mg of palbociclib once daily for 21 consecutive days

SUMMARY:
This is a one-site, interventional, prospective, single-arm, open-label, controlled phase-IIa trial evaluating the safety and efficacy of palbociclib in hospitalized, moderate COVID- 19 cases.

DETAILED DESCRIPTION:
The study will include hospitalized, moderate COVID-19 cases that have a risk of respiratory failure.

The study will generally consist of:

* A short screening phase (1 day) before enrollment and thus treatment decision.
* A 21 day treatment phase with one "cycle" of palbociclib
* An up to day 90 Safety Follow-Up Phase

The first three patients will be enrolled and treated one by one; the independent safety data review committee (ISRC) will review each patient after D21 before enrollment of the subsequent patient is permitted.

ELIGIBILITY:
Inclusion Criteria:

1. age >= 18 years
2. positive PCR COVID-19 test (max. 72h old)
3. known vaccination status
4. ANC >= 1,000/mm3 and platelets >= 50,000/mm3
5. willingness to participate (written informed consent)
6. established risk factors for a severe course of COVID-19-disease, for example: adipositas, cardiovascular disease including arterial hypertension, advanced age > 60, chronic lung disease including asthma, diabetis type I or II, chronic kidney disease, chronic liver disease
7. Oxygen supply: ≤ 2 liters/minute
8. Women of childbearing potential (WOCBP): must have a negative pregnancy test (ß- HCG urine or serum test) a. WOCBP is considered as i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile.

   b. Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.

   c. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.
9. Use of highly effective contraception method

   1. All potentially fertile participants, or their male partners, must use an adequate, medically approved method of contraception or agree to abstinence during and at least 3 weeks (females) and 14 weeks (males) after treatment with Palbociclib.
   2. For females, highly effective birth control should be used, i.e., combined hormonal contraception associated with inhibition of ovulation (oral, intravaginal, or transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, or implantable), intrauterine device, or intrauterine hormone-releasing system, bilateral tubal occlusion and vasectomized partner. As there is no information available on the interaction of palbociclib with oral contraceptives, a double-barrier contraception is necessary in this case.
   3. Males must agree to use a condom for at least 14 weeks after the treatment phase.

Exclusion Criteria:

1. age < 18 year
2. ECOG >= 3
3. ANC < 1,000/mm3 and platelets < 50,000/mm3
4. intensive care patient
5. treatment with any other CDK4/6 Inhibitor
6. pregnant or breast-feeding women
7. patients receiving immunosuppressants for other diseases (e.g. rheumatoid arthritis)
8. known malignancy in the past 5 years other than basal cell carcinoma
9. baseline O2-Saturation < 92%
10. participation in any other medical device or medicinal product study within the previous month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Rate of treatment-related treatment discontinuation after 21 days of palbociclib treatment | 21 days

SECONDARY OUTCOMES:
Time to freedom from oxygenation, measured in days after the first treatment dose. | 90 days
Time to transfer to ICU | 90 days
Course of neutrophil cell count during treatment | 21 days
Course of D-dimer during treatment | 21 days
Rate of thrombotic events during treatment | 21 days
Course of O2 saturation during treatment | 21 days
Rate of persisting symptoms after 3, 6, 9 and 12 months | Through completion of safety follow-up up to 12 month
Dose reduction rate | 21 days
Rate of (S)AEs at day 21 | at day 21

CONTACTS AND LOCATIONS:
Overall Officials: Mark Reinwald, PD Dr. med., Principal Investigator — Universitätsklinikum Brandenburg an der Havel
Locations (1):
- Universitätsklinikum Brandenburg an der Havel, Brandenburg, Germany